CLINICAL TRIAL: NCT04362410
Title: A Phase 1, Single Centre, Double-blind, Randomized, Placebo-controlled Parallel-group Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Immunogenicity of Tezepelumab After Single-Dose Subcutaneous Administration in Healthy Chinese Subjects (DIRECTION-CK)
Brief Title: Tezepelumab Phase 1 PK Study in Healthy Chinese Subjects
Acronym: DIRECTION-CK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00020
Record Dates: First submitted 2020-04-23; First posted 2020-04-24 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Safety; Tolerability; Immunogenicity; Tezepelumab; Healthy Chinese Subjects
MeSH Terms: interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: 48 healthy subjects will be randomly assigned to one of the three treatment cohorts (i.e. 1:1:1 to Low dose, Medium dose and High dose). 16 subjects will participate in each treatment cohort. Within each cohort, subjects will be randomized in a 3:1 ratio to receive a single dose of tezepelumab or placebo. Each subject will only participate in one cohort.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Tezepelumab: Low dose (Experimental): Tezepelumab: Tezepelumab single dose subcutaneously injection.
  Interventions: Biological: Experimental: Tezepelumab
- Tezepelumab: Medium dose (Experimental): Tezepelumab: Tezepelumab single dose subcutaneously injection.
  Interventions: Biological: Experimental: Tezepelumab
- Tezepelumab: High dose (Experimental): Tezepelumab: Tezepelumab single dose subcutaneously injection.
  Interventions: Biological: Experimental: Tezepelumab
- Placebo (Placebo Comparator): Placebo single dose subcutaneously injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Experimental: Tezepelumab — Tezepelumab single dose subcutaneously injection.
  Other Names: Tezepelumab
  Arms: Tezepelumab: High dose; Tezepelumab: Low dose; Tezepelumab: Medium dose
Other: Placebo — Placebo single dose subcutaneously injection.
  Arms: Placebo

SUMMARY:
This is a Phase 1, Single Centre, Double-blind, Randomized, Placebo-controlled Parallel-group Study to Evaluate the Pharmacokinetics, Safety, Tolerability and Immunogenicity of Tezepelumab after Single-Dose Subcutaneous Administration in Healthy Chinese Subjects.

DETAILED DESCRIPTION:
This is a Phase 1, single centre, randomized, double-blind, placebo-controlled, single dose, parallel group study in healthy Chinese male or female subjects. 48 healthy subjects will be randomly assigned to one of the three treatment cohorts (i.e. 1:1:1 to Low dose, Medium dose and High dose) to receive a single dose of tezepelumab or placebo in a 3:1 ratio. Each subject will only participate in one cohort. Dose level is unblinded and treatment (tezepelumab or placebo) will be double-blinded within each treatment cohort. Following a screening period of a maximum of 28 days, subjects will stay at the study facility for two nights starting from the day before dosing (Day -1) to Day 2. Subjects will receive a single dose of tezepelumab or placebo subcutaneously on Day 1 and safety monitoring and serial collection of blood samples for PK evaluation will be followed throughout the study period. The follow up period after the dosing will be 112 days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy Chinese subjects
* Age 18 to 45
* Body weight ≥ 40 kg
* Body mass index (BMI) between 19-24 kg/m2

Exclusion Criteria:

* History or evidence of a clinically significant disorder
* History of cancer
* Smokers of > 5 cigarettes/day
* Receipt of any marketed or investigational biologic within 4 months or 5 half-lives/non-biologic agent within 30 days or 5 half-lives prior to randomization
* History of chronic alcohol or drug abuse
* Hepatitis B, C or HIV
* Pregnant or breastfeeding
* History of anaphylaxis following any biologic therapy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

PRIMARY OUTCOMES:
AUC0-inf (Area under the serum concentration versus time curve from time zero to Infinity) | Blood samples will be collected from Day 1 (3 hour prior to administration of IP) and on Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85 and Day 113.
  To investigate the pharmacokinetics of single subcutaneous dose of tezepelumab in healthy Chinese subjects
AUC0-t (Area under the serum concentration versus time curve from time zero to the last quantifiable concentration) | Blood samples will be collected from Day 1 (3 hour prior to administration of IP) and on Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85 and Day 113.
  To investigate the pharmacokinetics of single subcutaneous dose of tezepelumab in healthy Chinese subjects
Cmax (Maximum serum concentration) | Blood samples will be collected from Day 1 (3 hour prior to administration of IP) and on Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85 and Day 113.
  To investigate the pharmacokinetics of single subcutaneous dose of tezepelumab in healthy Chinese subjects
tmax (time to Cmax) | Blood samples will be collected from Day 1 (3 hour prior to administration of IP) and on Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85 and Day 113.
  To investigate the pharmacokinetics of single subcutaneous dose of tezepelumab in healthy Chinese subjects
t1/2 (terminal serum half-life) | Blood samples will be collected from Day 1 (3 hour prior to administration of IP) and on Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85 and Day 113.
  To investigate the pharmacokinetics of single subcutaneous dose of tezepelumab in healthy Chinese subjects
CL/F (apparent serum clearance) | Blood samples will be collected from Day 1 (3 hour prior to administration of IP) and on Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85 and Day 113.
  To investigate the pharmacokinetics of single subcutaneous dose of tezepelumab in healthy Chinese subjects
Vz/F (apparent volume of distribution) | Blood samples will be collected from Day 1 (3 hour prior to administration of IP) and on Day 2, Day 4, Day 6, Day 8, Day 10, Day 12, Day 15, Day 22, Day 29, Day 43, Day 57, Day 85 and Day 113.
  To investigate the pharmacokinetics of single subcutaneous dose of tezepelumab in healthy Chinese subjects

SECONDARY OUTCOMES:
Immunogenicity anti-drug antibodies | Blood samples will be collected on Day 1 (3 hour prior to administration of IP) and on Day 29, Day 113.
  Incidence of anti-drug antibodies following single dose of tezepelumab

CONTACTS AND LOCATIONS:
Overall Officials: Jinfang Hu, Master, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- Research Site, Nanchang, China